CLINICAL TRIAL: NCT07357402
Title: Comparison of Clinical Outcomes, Parent and Child Satisfaction Between Stainless Steel Crowns and Prefabricated Hybrid (Bioflx) Crowns in Primary Molars
Brief Title: Clinical Outcomes and Satisfaction of Stainless Steel vs Bioflx Crowns in Primary Molars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PHAM LE ANH THY (Other)
Responsible Party: Sponsor-Investigator, PHAM LE ANH THY, Dentist, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3526/QĐ-ĐHYD
Record Dates: First submitted 2026-01-17; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Severely Decayed Primary Molars Requiring Full-Coverage Crowns
Keywords: Stainless steel crowns; Bioflx crowns; Primary molars; Split-mouth study; Parental and child satisfaction

STUDY DESIGN:
Intervention Model Description: The study is designed as a randomized split-mouth clinical trial. Each child will receive both types of crowns on two similar teeth on opposite sides of the mouth. One side is randomly assigned to receive a stainless steel crown, and the other side receives a Bioflx crown. The placement of the two crowns is performed in two separate appointments, with an interval of 1 to 2 weeks between them. This approach allows the child to adapt to the new occlusion (bite) after the first crown is placed, ensuring a more stable result before the second procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Stainless steel crown (Active Comparator): Participants receive a prefabricated stainless steel crown placed on a primary molar according to standard pediatric dental procedures. The crown is selected, adapted, and cemented following conventional clinical protocols and serves as the standard treatment comparator in this study.
  Interventions: Device: Stainless Steel Crown
- Bioflx crown (Experimental): Participants receive a prefabricated Bioflx crown placed on a primary molar using manufacturer-recommended techniques. The crown is selected and cemented following standardized clinical procedures and is evaluated as the experimental intervention for clinical performance and patient-related outcomes.
  Interventions: Device: Bioflx crown

INTERVENTIONS:
Device: Stainless Steel Crown — Stainless steel crowns are prefabricated metal crowns that have been widely and long used in pediatric dentistry to restore primary molars with extensive caries or following pulp therapy.
  Arms: Stainless steel crown
Device: Bioflx crown — Bioflx crowns are prefabricated tooth-colored polymer crowns designed to improve esthetics compared with conventional stainless steel crowns
  Arms: Bioflx crown

SUMMARY:
The goal of this clinical trial is to learn if the Bioflx crown (a tooth-colored material) is as effective as the standard stainless steel crown for treating severely decayed baby back teeth in children aged 4 to 10 years old. The study also aims to evaluate parent and child satisfaction with these restorative options.

The main questions it aims to answer are:

1. Is the Bioflx crown as effective as the stainless steel crown in terms of durability, staying in place, and protecting the tooth from new decay?
2. Does the Bioflx crown maintain better gum health and cause less wear on the opposing teeth compared to the stainless steel crown?

Researchers will compare the Bioflx crown to the stainless steel crown to see which material works better to restore tooth function and health.

Participants will:

1. Receive one Bioflx crown and one stainless steel crown on similar teeth on opposite sides of the mouth.
2. Visit the clinic for two separate appointments, spaced 1 to 2 weeks apart, to have the crowns placed.
3. Return for checkups at 3 months and 6 months so researchers can examine the health of the teeth and gums.
4. Answer questions about how happy they are with the appearance and feel of the crowns.

DETAILED DESCRIPTION:
The standard treatment for fixing severely decayed baby back teeth is the stainless steel crown, which is a durable metal cap. While these metal crowns work very well, many parents and children prefer a more natural, tooth-colored look. This study tests a newer option called the Bioflx crown, which is made of a flexible, tooth-colored material.

The Treatment Process The crowns are placed during two separate visits, usually 1 to 2 weeks apart. It gives the child time to get used to the first crown and ensures their bite is comfortable before the second one is placed. It makes the appointments shorter and easier for the child to handle. The side of the mouth that gets the metal crown and the side that gets the tooth-colored crown is randomized.

How Success is Measured

After the crowns are placed, researchers will check them again at 3 months and 6 months. They will use professional standards to evaluate the effectiveness of the crowns, focusing on:

1. Durability: Do the crowns stay glued to the teeth and resist wearing down from chewing?
2. Prevention: Does the new material prevent new cavities from forming at the edges of the crown?
3. Gum Health: Do the gums around the tooth stay healthy, or do they become red and swollen?
4. Satisfaction: How do the child and parent feel about the color, size, and shape of the tooth-colored crown compared to the metal one?

ELIGIBILITY:
Inclusion Criteria:

* Children with at least two carious primary molars located on both the right and left sides of the dental arch and indicated for crown placement
* Children and their parents have ability to communicate in Vietnamese
* Primary molars indicated for full-coverage crown restoration, including teeth with:

  * Multi-surface caries
  * Extensive caries or enamel-dentin defects
  * Interproximal caries
  * High risk of failure with other restorative materials
  * Teeth following pulpotomy or pulpectomy

Exclusion Criteria:

* Uncooperative children
* Presence of psychiatric or neurological disorders affecting communication ability
* Malocclusion (crossbite or scissors bite)
* Having abnormal parafunctional habits
* Teeth with root resorption exceeding one half of the root length

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
- Clincal outcomes: crown stability; bite discomfort; fit and color changes at the crown edge; crown shape; crown retention; crown wear; wear of the opposing tooth or crown - Oral hygiene and gum health around the crowns | - Crown stability, bite discomfort, fit and color at the crown margin, and crown shape were checked after crown placement, at 3 months, and at 6 months follow-up visits. Others were checked at 3, 6 months, except secondary caries was checked at 6 months
  * Each clinical parameter was assessed using the modified United States Public Health Service (USPHS) criteria.
    * Outcomes were rated on a three-level scale (Alpha, Bravo, Charlie), where Alpha indicates an ideal condition, Bravo an acceptable condition with minor defects, and Charlie an unacceptable condition requiring repair or replacement. For analysis, Alpha and Bravo scores were considered acceptable, while Charlie scores were considered failures.
    * Secondary caries were assessed using periapical radiographs, while all other clinical parameters were assessed by dental explorer and documented using photographs (Canon 6D camera).
  * This outcome evaluates how clean the teeth are and how healthy the gums are around crowned teeth. Plaque and gum condition were evaluated using standard dental indices (Plaque Index and Gingival Index). Dentists exam by using a periodontal probe at six points around the crowns, and the scores were combined to provide an overall result.

SECONDARY OUTCOMES:
parent and child satisfaction | From immediately after crowns placement through the 3-month and 6-month follow-up visits.
  * Children's and parents' satisfaction are assessed using two separate questionnaires, both employing a 5-point Likert scale with scores ranging from 1 to 5 (Units on a Scale). For children, a facial expression Likert scale is used.
  * The Likert scale levels are defined as follows:
    1. - Very dissatisfied
    2. - Dissatisfied
    3. - Neutral
    4. - Satisfied
    5. - Very satisfied
  * Higher scores indicate greater satisfaction
  * Parent questionnaire includes the following items: size, shape, color of two crowns; child's ability to eat a variety of foods after treatment and overall parental satisfaction.
  * Another questionnaire scale based on children ratings of treatment on them consists of five categories, including 1) Appearance of the teeth before crown placement; 2) Crowns have improved the appearance of the child's teeth; 3) The child avoided smiling before crowns; 4) Child smiling after crowns; 5) The oral health of the child improved after crowns.

CONTACTS AND LOCATIONS:
Overall Officials: Huong Thi Nguyen Nguyen, PhD, Study Chair — Faculty of Dentistry, University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tin BT, Phuong NTM, Anh NTH, Bau TH, Dong TT, Ngoc VTN. Short-Term Clinical Evaluation of Bioflx Crowns for Primary Molar Restoration in Children Aged 4-8 Years in Vietnam: A Pilot Observational Study. Int J Paediatr Dent. 2026 Jan;36(1):187-194. doi: 10.1111/ipd.70039. Epub 2025 Oct 22. PMID 41126408
- [Background] Klabunde RE, Althouse DG. Adenosine metabolism in dog whole blood: effects of dipyridamole. Life Sci. 1981 Jun 8;28(23):2631-41. doi: 10.1016/0024-3205(81)90721-9. No abstract available. PMID 7266243
- [Background] Lopez-Cazaux S, Aiem E, Velly AM, Muller-Bolla M. Preformed pediatric zirconia crown versus preformed pediatric metal crown: study protocol for a randomized clinical trial. Trials. 2019 Aug 24;20(1):530. doi: 10.1186/s13063-019-3559-1. PMID 31445509
- [Background] Pozos-Guillen A, Chavarria-Bolanos D, Garrocho-Rangel A. Split-mouth design in Paediatric Dentistry clinical trials. Eur J Paediatr Dent. 2017 Mar;18(1):61-65. doi: 10.23804/ejpd.2017.18.01.13. PMID 28494606
- [Background] Patil AS, Jain M, Choubey S, Patil M, Chunawala Y. Comparative evaluation of clinical success of Stainless Steel and Bioflx crowns in primary molar - A 12 month split mouth prospective randomized clinical trial. J Indian Soc Pedod Prev Dent. 2024 Jan 1;42(1):37-45. doi: 10.4103/JISPPD.JISPPD_484_23. Epub 2024 Apr 15. PMID 38616425